CLINICAL TRIAL: NCT03021863
Title: How Frequently and in What Format Are Research Trial Results Disseminated to Participants? A Survey of Trialists and Response Questionnaire Trial
Brief Title: How Frequently and in What Format Are Research Trial Results Disseminated to Participants (ResponseQT)
Acronym: ResponseQT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ThinkWell (Other)
Collaborators: University of Oxford (Other); The BMJ (Other); Queen's University, Belfast (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: ThinkWell & BMJ 2
Record Dates: First submitted 2017-01-11; First posted 2017-01-16 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Motivation
Keywords: Dissemination; Tone; Survey reminders; Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- Group A Reminder (Active Comparator): Tone of reminder email (duty 14 days followed by duty for non-responders 28 days)
  Interventions: Behavioral: Group A Reminder
- Group B Reminder (Active Comparator): Tone of reminder email (encouragement 14 days followed by encouragement for non-responders 28 days)
  Interventions: Behavioral: Group B Reminder
- Group C Reminder (Active Comparator): Tone of reminder email (encouragement 14 days followed by duty for non-responders 28 days)
  Interventions: Behavioral: Group C Reminder
- Group D Reminder (Active Comparator): Tone of reminder email (duty 14 days followed by encouragement for non-responders 28 days)
  Interventions: Behavioral: Group D Reminder
- Group E Reminder (Active Comparator): Tone of reminder email (generic reminders at 14 days followed by generic for non-responders 28 days)
  Interventions: Behavioral: Group E Reminder
- Group F Reminder (Active Comparator): Tone of reminder email (generic 14 days followed by duty for non-responders 28 days)
  Interventions: Behavioral: Group F Reminder
- Group G Reminder (Active Comparator): Tone of reminder email (generic 14 days followed by encouragement for non-responders 28 days)
  Interventions: Behavioral: Group G Reminder
- Group H Reminder (Active Comparator): Tone of reminder email (duty 14 days followed by generic for non-responders 28 days)
  Interventions: Behavioral: Group H Reminder
- Group I Reminder (Active Comparator): Tone of reminder email (encouragement 14 days followed by generic for non-responders 28 days)
  Interventions: Behavioral: Group I Reminder

INTERVENTIONS:
Behavioral: Group A Reminder — Tone of reminder email (duty 14 days followed by duty 28 days for non-responders)
  Arms: Group A Reminder
Behavioral: Group B Reminder — Tone of reminder email (encouragement 14 days followed by encouragement 28 days for non-responders)
  Arms: Group B Reminder
Behavioral: Group C Reminder — Tone of reminder email (encouragement 14 days followed by duty for non-responders 28 days)
  Arms: Group C Reminder
Behavioral: Group D Reminder — Tone of reminder email (duty 14 days followed by encouragement for non-responders 28 days)
  Arms: Group D Reminder
Behavioral: Group E Reminder — Tone of reminder email (generic reminders 14 days followed by 28 days for non-responders)
  Arms: Group E Reminder
Behavioral: Group F Reminder — Tone of reminder email (generic 14 days followed by duty for non-responders 28 days)
  Arms: Group F Reminder
Behavioral: Group G Reminder — Tone of reminder email (generic 14 days followed by encouragement for non-responders 28 days)
  Arms: Group G Reminder
Behavioral: Group H Reminder — Tone of reminder email ( duty14 days followed by generic for non-responders 28 days)
  Arms: Group H Reminder
Behavioral: Group I Reminder — Tone of reminder email (encouragement 14 days followed by generic non-responders 28 days)
  Arms: Group I Reminder

SUMMARY:
Questionnaires are frequently used in online research, however recruiting, and completion rates of online participants from a variety of cultures and demographic backgrounds can be challenging. The challenge is greater in an online cohort because there is no way to observe the participant beyond what is contributed online. Poor recruiting and completion can result in underpowered research that may not be representative of the sample population. This can trigger an increase in costs as the recruitment period may have to be extended until sample size is reached. When recruiting and completion rates are inadequate studies may have to be terminated and the answer to the research question can remain unknown.

To mitigate these challenges, reminder emails are sent to questionnaire respondents. There is uncertainty about how the tone of the email reminder affects the proportion of recruitment rates.

A nested randomized trial will be used to test the intervention of tone delivery in survey email reminders to establish an evidence base. This study (ResponseQT) proposes to link with the anticipated 20,000 person international cohort study, (How Frequently and in What Format are Research Trial Results Disseminated to Participants: A Survey of Trialists (ResponseQT) to explore the evidence of effect for the research question, "Does the tone of a survey email reminder affect the proportion of survey participants recruited. The population will consist of researchers who have published a clinical trial indexed in Pub Med in 2014-15.The intervention is the tone of questionnaire email reminders and the outcomes will be the proportion of participants recruited after invitation (partial plus complete responses) following reminder 1 and 2.

DETAILED DESCRIPTION:
RATIONALE

Dissemination is the planned process by which results of studies are communicated to the stakeholders of that research. Stakeholders can include health policy makers, academics, practicing clinicians and other health service workers, patients, the general public, and research funders. There are multiple ways to disseminate research findings and it is often considered a shared responsibility between funders and research investigators. Traditionally, the focus has targeted healthcare professionals, policy makers, and academics through journal publications and conference presentations. However, optimal knowledge translation depends on disseminating results to all stakeholders in a way that enables them to consider the implications of the results.

Effective communication and active dissemination of research results to patients and the lay public is essential for making informed decisions and choices, but it is sometimes considered as an afterthought. Furthermore, there is no consensus on what dissemination to patients or members of the lay public means, what is the most effective dissemination process and whether research results should be disseminated to relevant patient groups and the wider public as well as the patients who took part in the studies.

Only clinical trials indexed in PubMed 2014-15 where participants were enrolled into the study will be included. We will include screening questions at the start of the survey to exclude authors of non-randomised controlled trials, preclinical, and first-in-human trials and trials where there were no study participants.

AIM

To identify frequency and format of dissemination of clinical trial results to participants and to identify barriers to dissemination.

OBJECTIVES

1. To identify frequency of dissemination of recently published clinical trial results to participants;
2. To explore the format of results disseminated to participants and describe researchers' perceived appropriateness and accessibility of the format;
3. To identify how frequently research results are disseminated to patients beyond those taking part in the trials such as via advocacy groups;
4. To explore the frequency of public/patient involvement for determining the format, content, and extent of the dissemination plans;
5. To determine researchers' perceived confidence in disseminating results to participants and other patients.

This research will contain a study within a study (SWAT) also known as a nested trial (ResponseQT).

SWAT RATIONALE

Written communication in questionnaire email reminders are without verbal or sensory cues and it is difficult to modify reminders without feedback from respondents. It would be helpful to know what kind of tone the researcher can take to increase recruitment rates.

In questionnaires, the tone could be perceived as the perception of the researcher's attitude toward the reader and the subject of the message. The overall tone of a questionnaire reminder message may affect the reader just as one's tone of voice affects the listener in a verbal exchange. This could influence response and completion rates. Added to the complexity, tone can be interpreted differently by different individuals. Survey communications about reminders suggest two approaches appealing to a team victory with a sense of duty and benefit for others by participating or by building a sense of encouragement for participation. In addition, we will test whether introducing duty or encouragement in the second reminder (after a generic first reminder) makes a difference and whether someone who was exposed to duty or encouragement in the first reminder benefits from the reinforcement of a "nudge" from a generic reminder.

METHODS

This research involves exploring ways to increase recruitment rates through reminder emails that will be sent to those who were invited but have not yet responded to the questionnaire. A reminder will be sent to all non-respondents by email 14 days following the initial mailing. An additional reminder will be sent to all non-respondents by email 28 days following the first reminder. The nested trial (ResponseQT) will examine the evidence of effect for tone used within the questionnaire reminder emails. The group to which a participant is randomized will determine the tone of the questionnaire reminder emails.

All potential respondents will be randomized to one of nine groups. They will receive the same questionnaire invitation email. Reminders for non-responders be assigned according to the group they were randomized to:

Group A Tone = Duty x 2

Group B Tone = Encourage x 2

Group C Tone = Encourage + Duty

Group D Tone = Duty + encourage

Group E Tone = Generic tone reminders X 2

Group F Tone = Generic + Duty

Group G Tone = Generic + Encouragement

Group H Tone = Duty + Generic

Group I Tone = Encouragement + Generic

All non-responders will receive a reminder to complete the questionnaire at fourteen days according to the group they are randomized to. At twenty-eight days remaining non-responders will receive the second reminder email.

The outcomes of recruitment will be compared at three stages: initial response, following the first reminder and following the second reminder.

ELIGIBILITY:
Inclusion Criteria:

* reports of clinical trials with human participants indexed in PubMed 2014-15

Exclusion Criteria:

* reports of laboratory or animal studies,
* reports of preclinical trials,
* reports of trials where there were no study participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1198 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Recruitment | Duration of study up to 60 days
  Proportion of sample recruited

CONTACTS AND LOCATIONS:
Overall Officials: Amy I Price, PhD, Principal Investigator — ThinkWell
Locations (1):
- ThinkWell, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-Identified, aggregated data upon request to investigators due to data protection laws

REFERENCES:
- [Background] Wilson PM, Petticrew M, Calnan MW, Nazareth I. Disseminating research findings: what should researchers do? A systematic scoping review of conceptual frameworks. Implement Sci. 2010 Nov 22;5:91. doi: 10.1186/1748-5908-5-91. PMID 21092164
- [Background] Tetroe JM, Graham ID, Foy R, Robinson N, Eccles MP, Wensing M, Durieux P, Legare F, Nielson CP, Adily A, Ward JE, Porter C, Shea B, Grimshaw JM. Health research funding agencies' support and promotion of knowledge translation: an international study. Milbank Q. 2008 Mar;86(1):125-55. doi: 10.1111/j.1468-0009.2007.00515.x. PMID 18307479
- [Background] Felix LM, Burchett HE, Edwards PJ. Factorial trial found mixed evidence of effects of pre-notification and pleading on response to Web-based survey. J Clin Epidemiol. 2011 May;64(5):531-6. doi: 10.1016/j.jclinepi.2010.06.001. Epub 2010 Sep 17. PMID 20850270
- [Background] Fang J, Shao P, Lan G. Effects of innovativeness and trust on web survey participation. Comput Human Behav 2009;25:144-52. doi:10.1016/j.chb.2008.08.002
- [Background] Fan W, Yan Z. Factors affecting response rates of the web survey: A systematic review. Comput Human Behav 2010;26:132-9. doi:10.1016/j.chb.2009.10.015
- [Background] Cook DA, Wittich CM, Daniels WL, West CP, Harris AM, Beebe TJ. Incentive and Reminder Strategies to Improve Response Rate for Internet-Based Physician Surveys: A Randomized Experiment. J Med Internet Res. 2016 Sep 16;18(9):e244. doi: 10.2196/jmir.6318. PMID 27637296
- [Background] Baruch Y, Holtom BC. Survey response rate levels and trends in organizational research. Hum Relations 2008;61:1139-60. doi:10.1177/0018726708094863